CLINICAL TRIAL: NCT04565145
Title: A Phased Clinical Trial of a Dietary Supplement Kava: Biomarker Changes and Anxiolytic Effects Phase 2: Kava Biomarker
Brief Title: Biomarker Changes and Anxiolytic Effects-Phase 2
Acronym: KavaPK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Thorne HealthTech, Inc (Industry); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB202001129 -A; IRB201900074-N (Other: UF IRB (Phase I)); 1R61AT009988-01A1 (NIH); OCR36443 (Other: UF OnCore); 3R61AT009988-02S1 (NIH)
Record Dates: First submitted 2020-09-14; First posted 2020-09-25 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: Pharmacokinetics
Keywords: kava; dietary supplement; anxiety; generalized anxiety disorder (GAD)
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Kava Pharmacokinetics Group (Experimental): 75 mg kava dietary supplement capsules per day for one week.
  Interventions: Drug: Kava Dietary Supplement
- Placebo (Placebo Comparator): Three placebo capsule per day for one week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Kava Dietary Supplement — Participants will be given three 75mg kava capsules per day for one week
  Other Names: Flavokavain AB-free kava
  Arms: Kava Pharmacokinetics Group
Drug: Placebo — Participants will be given three placebo capsules per day for one week
  Arms: Placebo

SUMMARY:
This study will examine the utility of plasma and urinary based biomarkers for the anxiolytic properties of kava. The investigators will conduct a one week, double blind, randomized placebo controlled trial of kava, dosed at three 75 mg capsules per day, vs placebo, in adults with generalized anxiety disorder.

DETAILED DESCRIPTION:
This study will examine the utility of plasma and urinary based biomarkers for the anxiolytic properties of kava, a natural dietary supplement. The investigators will conduct a one week, double blind, randomized placebo controlled trial of kava, dosed at three 75 mg capsules per day, vs placebo, in adults with generalized anxiety disorder. Clinical measures of anxiety, blood, and urine will be obtained. Biomarkers of interest include PRKACA, cortisol, urinary TCE, and NA5HT. Participants will be assessed pre- and post-treatment. The participants will also be followed for 12 weeks after the end of treatment to identify any potential rare adverse events, particularly liver toxicity, that appear in a delayed fashion.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-50 who meet Diagnostic Statistical Manual (DSM)-5 criteria for GAD as the primary psychiatric diagnosis
* No more than one failed therapeutic trial of an FDA approved medication for the treatment of GAD
* Score of>14 on the Hamilton Anxiety Rating Scale at both screening and baseline
* At least a 4 (moderate) on the Clinical Global Impressions Severity Scale at both screening and baseline
* Females of potential childbearing status must use adequate contraceptive precautions.

Exclusion Criteria:

* Unwilling/unable/unsafe to stop psychotropic medications (if on any) for the duration of the study
* Inability to refrain from acetaminophen, alcohol or other potentially hepatotoxic substances
* History of liver disease or current liver disease or clinically significant elevation in serum liver chemistries
* Unstable medical or neurological condition
* Positive urine drug screen for substances of abuse
* Active substance abuse/dependence
* Lifetime history of a psychotic disorder, bipolar disorder, PTSD or Obsessive Compulsive Disorder
* Any significant risk for self-harm or suicidality as determined by the principal investigator or suicide attempt within the last 6 months
* Psychotherapy newly instituted during the 6 weeks leading up to enrollment in the study. Subjects established in psychotherapy without change during the course of the study may participate
* Montgomery-Asberg Depression Rating Scale (MADRS) > 17 (moderate or severe depressive symptoms)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Mathews, MD, Principal Investigator — University of Florida
Locations (1):
- UF CTSI Clinical Research Center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals were recruited from flyers that were distributed in and around the Gainesville area and from the University of Florida (UF) Psychiatry and Psychology clinics.
Pre-assignment Details: Individuals were excluded it the met any of the exclusion criteria at screening or baseline.
Period: Overall Study
Arm/Group | Kava Pharmacokinetics Group | Placebo
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Participants were enrolled and analyzed as described in the protocol
Groups:
- Total: Total of all reporting groups
Arm/Group | Kava Pharmacokinetics Group | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 26 [19 to 50] | 23 [18 to 37] | 25 [18 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 9 | 7 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 9 | 7 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Mean PRKACA Change
Description: The change in mean PRKACA value from pre to post-treatment
Time Frame: From Baseline (pre dose) to 1 week after taking the first dose (post dose)
Measure: Mean (Standard Deviation); unit: relative fluorescence units
Arm/Group | Kava Pharmacokinetics Group | Placebo
Number analyzed (Participants) | 10 | 10
relative fluorescence units
  Pre dose PRKACA | 7224.56 (3526.22) | 5348.93 (2027.02)
  Post dose PRKACA | 6307.21 (5887.36) | 6495.7 (3757.65)

ADVERSE EVENTS:
Time Frame: 1 year and 6 months
Description: Guidelines for reporting adverse events were the same as the clinical trials.gov definition.
Arm/Group | Kava Pharmacokinetics Group | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 4/10 | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Kava Pharmacokinetics Group (N=10) | Placebo (N=10)
Headache (General disorders) | 2 (2) | 1 (1) — Headache
Dizziness (General disorders) | 1 (1) | 1 (1) — Dizziness
Appetite loss (General disorders) | 1 (1) | 1 (1) — Appetite loss
Fatigue (General disorders) | 2 (2) | 0 (0) — Fatigue
Chest tightness (General disorders) | 0 (0) | 1 (1) — Chest tightness
Brain fog (General disorders) | 0 (0) | 1 (1) — Brain fog
Vivid dreams (General disorders) | 0 (0) | 1 (1) — Vivid dreams

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT04565145/Prot_SAP_001.pdf
  • Informed Consent Form (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/45/NCT04565145/ICF_000.pdf